CLINICAL TRIAL: NCT05147844
Title: Antitumor Activity of Toripalimab Combined With Radiotherapy in the Treatment of Oligometastatic Nasopharyngeal Carcinoma: A Single-arm, Multicenter Study
Brief Title: Toripalimab Combined With Radiotherapy in the Treatment of Oligometastatic Nasopharyngeal Carcinoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Xinqiao Hospital of Chongqing (Other)
Collaborators: Southwest Hospital, China (Other); Daping Hospital and the Research Institute of Surgery of the Third Military Medical University (Other); Chongqing University Cancer Hospital (Other)
Responsible Party: Principal Investigator, Jianguo Sun, director physician, Xinqiao Hospital of Chongqing
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XQonc-017
Record Dates: First submitted 2021-11-23; First posted 2021-12-07 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Nasopharyngeal Carcinoma
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — toripalimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Toripalimab +Radiotherapy (Experimental)
  Interventions: Drug: Toripalimab

INTERVENTIONS:
Drug: Toripalimab — Toripalimab: 240mg, iv. Q3W for 1 year or until disease progression/intolerable toxicity
  Radiotherapy:
  Newly diagnosed patients: IMRT for nasopharynx lesions and cervical lymph nodes, pGTVnx 70 Gy, pGTVnd 99Gy, pCTV1, 60 Gy, pCTV2, 54 Gy, 33 times, completed in 7 weeks.
  Relapsed patients: IMRT for nasopharynx lesions and cervical lymph nodes, pGTVnx 60Gy, pGTVnd 60Gy, 20-25 times, completed in 4-5 weeks.
  Newly diagnosed and relapsed patients: SBRT for oligometastatic lesions, pGTV 25-40 Gy, 3-5 times, completed in 1-2 weeks.
  Other Names: JS001

SUMMARY:
The aim of the study was to determine the efficacy and safety of toripalimab combined with radiotherapy in the treatment of oligometastatic nasopharyngeal carcinoma

DETAILED DESCRIPTION:
Chemotherapy has been widely used for the treatment of relapsed or metastatic nasopharyngeal carcinoma. However, the long-term survival and quality of life of patients was still unsatisfactory. In this prospective, multicenter, single arm study, the efficacy and safety of toripalimab combined with radiotherapy in the treatment of oligometastatic nasopharyngeal carcinoma is determined.

ELIGIBILITY:
Inclusion Criteria:

1. Must have signed written informed consent and able to comply with study procedure
2. 18-75 years old
3. Histologically or cytologically confirmed nasopharyngeal carcinoma
4. Pathology or imaging confirmed metastatic nasopharyngeal carcinoma.( Clinical stage of IVB according to the 8th edition of AJCC)
5. Imaging (preferred PET-CT) confirmed oligometastatic NPC (defined as ≤5 metastatic lesions, ≤2 metastatic organs)
6. Have not received any treatment for metastatic nasopharyngeal carcinoma.
7. Unsuitable or unwilling to receive chemotherapy according to the judgment of investigator.
8. Eastern Cooperative Oncology Group (ECOG) Performance Status score 0-1
9. Estimated life ≥ 6 month
10. At least 1 measurable lesions according to RECIST v1.1
11. Adequate organ function, defined as achieving the following laboratory test results within 7 days before enrollment: ANC≥1.5×10^9/L，PLT≥100×10^9/L，Hb≥90g/L((Have not accepted blood transfusion or growth factors within 14 days)；the international normalized ratio (INR) or prothrombin time (PT) ≤ 1.5 × ULN; activated partial thromboplastin time(APTT) ≤1.5 × ULN；serum creatinine≤1.5×ULN or estimated glomerular filtration rate(GFR) ≥ 60 mL/min/1.73 m2; total bilirubin≤1.5×ULN（total bilirubin<3×ULN for patients with Gilbert syndrome）; AST and ALT ≤ 2.5×ULN (AST and ALT ≤ 2.5×ULN for patients with liver metastasis);

Exclusion Criteria:

1. Allergy to any component of toripalimab
2. With any active autoimmune disease or a history of autoimmune disease that may relapse

   Note: Patients with the following diseases were not excluded and should be further screened:

   Controlled type 1 diabetes; Hypothyroidism (could be controlled just by hormone replacement therapy); Controlled celiac disease; Skin diseases that do not require systemic treatment (e.g. vitiligo, psoriasis, alopecia); Any other disease which is not expected to be relapsed without external stimulate
3. Any active malignancy ≤ 2 years before randomization except for the specific cancer under investigation in this study and any locally relapsed cancer that has been cured after treatment (eg, resected basal or squamous cell skin cancer, superficial bladder cancer, carcinoma in situ of the cervix or breast)
4. Received corticosteroid therapy at a dose ≥ 10 mg prednisone per day or any other systemic immunosuppressive therapy within 14 days prior to enrollment.
5. Patient with uncontrolled diabetes, or abnormal potassium, sodium or corrected calcium levels (≥ grade 1) after receiving standard treatment, or ≥ grade 3 hypoalbuminemia within 14 days prior to enrollment
6. Patient with a history of interstitial lung disease, non-infectious pneumonia or uncontrollable diseases, including pulmonary fibrosis, acute lung disease, hypertension, etc.
7. Evidence of severe chronic or active infections (including tuberculosis infection) requiring systemic antibiotics, antibacterial or antiviral therapy within 14 days prior to enrollment
8. Patient with a history of HIV infection
9. Evidence of contraindications of immunotherapy or radiotherapy
10. Patient with untreated chronic hepatitis B or HBV-DNA≥ 500 IU/mL, or active hepatitis C.

    Note: Patients with inactive infection of hepatitis B surface antigen (HBsAg), stable hepatitis B after treatment (HBV DNA < 500 IU/mL）and cured hepatitis C could be included.
11. Have undergone any operation requiring general anesthesia within 28 days prior to enrollment
12. Previous allogeneic stem cell transplantation or organ transplantation
13. Patient with any of the following cardiovascular risk factors: Cardiogenic chest pain within 28 days prior to enrollment, which is defined as moderate pain that limits instrumental activities of daily life; Symptomatic pulmonary embolism within 28 days prior to enrollment; Acute myocardial infarction within 6 months prior to enrollment; Grade III or IV disease according to the New York Heart Association within 6 months prior to enrollment;≥ Grade 2 ventricular arrhythmias within 6 months prior to enrollment or the first administration; With a history of cerebrovascular accident within 6 months prior to enrollment or the first administration
14. Grade 2 peripheral nerve disease according to NCI-CTCAE V5.0
15. Underlying medical conditions (including abnormal laboratory test values) that: affect drug administration; affect the interpretation of toxicity or AE; lead to poor compliance; alcohol or drug abuse or dependence
16. Participate in another interventional clinical study at the same time

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
1-year progression-free survival rate according to RECIST v1.1 | From date of randomization, until disease progression , loss of clinical benefit ,withdrawal of consent, death, or study termination by the Sponsor, whichever occurs first. 1 year
  To evaluate the efficacy of Toripalimab plus radiotherapy in patients with oligometastatic nasopharyngeal carcinoma, as measured by 1-year progression-free survival rate according to RECIST v1.1

SECONDARY OUTCOMES:
PFS according to RECIST v1.1 | From date of randomization, until disease progression , loss of clinical benefit ,withdrawal of consent, death, or study termination by the Sponsor, whichever occurs first. Up to 2 approximately years
  To evaluate the efficacy of Toripalimab plus radiotherapy in patients with oligometastatic nasopharyngeal carcinoma, as measured by progression-free survival rate according to RECIST v1.1
OS | up to 5 years
  To evaluate the efficacy of Toripalimab plus radiotherapy in patients with oligometastatic nasopharyngeal carcinoma, as measured by overall survival (OS)
2-year progression-free survival rate according to RECIST v1.1 | From date of randomization, until disease progression , loss of clinical benefit ,withdrawal of consent, death, or study termination by the Sponsor, whichever occurs first. Up to 2 approximately years
  To evaluate the PFS rate at 2 years in the treatment arm
2-year overall survival | From date of randomization until death, loss to follow-up, or study termination by the Sponsor whichever occurs first.Up to 3.5 approximately years
  To evaluate the OS rate at 2 years in the treatment arm
1-year progression-free survival rate according to irRECIST | From date of randomization, until disease progression , loss of clinical benefit ,withdrawal of consent, death, or study termination by the Sponsor, whichever occurs first. Up to 1 approximately year
  To evaluate the efficacy of Toripalimab plus radiotherapy in patients with oligometastatic nasopharyngeal carcinoma, as measured by 1-year progression-free survival rate according to irRECIST
ORR according to RECIST v1.1 | From date of randomization, until disease progression , loss of clinical benefit ,withdrawal of consent, death, or study termination by the Sponsor, whichever occurs first. Up to 2 approximately years
  To evaluate the efficacy of Toripalimab plus radiotherapy in patients with oligometastatic nasopharyngeal carcinoma, as measured by investigator-assessed overall response rate (ORR) according to RECIST v1.1.
DCR according to RECIST v1.1 | From date of consent informed until 60 days after the last investigational product administration. Up to 2 approximately years
  To evaluate the efficacy of Toripalimab plus radiotherapy in patients with oligometastatic nasopharyngeal carcinoma, as measured by investigator-assessed disease control rate (DCR) according to RECIST v1.1
DoR according to RECIST v1.1 | From date of randomization, until disease progression , loss of clinical benefit ,withdrawal of consent, death, or study termination by the Sponsor, whichever occurs first. Up to 2 approximately years
  To evaluate the efficacy of Toripalimab plus radiotherapy in patients with oligometastatic nasopharyngeal carcinoma, as measured by investigator-assessed duration of response (DoR) according to RECIST v1.1
AE(SAE) | From date of consent informed until 60 days after the last investigational product administration. Up to 2 approximately years
  Incidence of serious adverse events(SAE) as assessed by CTCAE version 5.0

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Xinqiao Hospital of Chongqing, Chongqing, Chongqing Municipality
  - the second affiliated hospital of Army medical university, Chongqing, Chongqing Municipality

IPD SHARING:
Plan to Share IPD: No